CLINICAL TRIAL: NCT06721637
Title: Effect of Core Stability Exercise Versus Whole Body Vibration in Improving Vitamin D Absorption in Women
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, Assistant professor of physical therapy, October 6 University
Other Study IDs: IRB#18\11\2024-2025
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Vitamin D Absorption
Keywords: Core stability exercise; Whole body vibration; Vitamin D absorption; Women

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (n = 20): received core stability exercise trained three times a week for 8 weeks.: 1. Abdominal hollowing exercise:
     Woman was in crook lying position with feet flat on the treatment table. The therapist put his two thumbs on the anterior superior iliac spines then, asked the woman to contract the abdominal muscle, hold the contraction for 10 seconds, then, asked her to relax for 10 seconds [29].
  2. Quadruped abdominal hollowing exercise:
     Woman was in a quadruped position on the treatment plinth with her hips, knees and shoulders flexed 90 degrees, the spine parallal to the table. The woman instructed to inhale allowing her abdomen to drop, as she exhale, she was pulling her abdominal toward her spine without moving her spine with holding for 10 seconds while maintaining her normal breathing patterns. Then asked the woman to relax for 10 seconds [29].
  3. Bilateral knee raise exercise:
  Woman was in crook lying position .She instructed to contract her lower abdomen while continuing to breathe in a normally. While maintaining the contraction
  Interventions: Combination Product: Group A (n = 20): received core stability exercise trained three times a week for 8 weeks.
- Group B (n = 20): received whole body vibration trained three times a week for 8 weeks: The woman assumed a full squat position on a vibration platform. The apparatus was set at a frequency of 30 Hz, amplitude of 2 mm, and duration of 5 min. The women were instructed to remain in the squatting position with holding hand rail after turning on the vibration and to report any discomfort that might arise. At the end of 5 min, the vibration turned off automatically. Thereafter, the women took a 1-min rest. They were then asked to stand on the vibration platform for 5 min, with the same parameters as those used in the squatting position. Thus, the total time for the application of WBV in each session was 10 min
  Interventions: Device: Group B (n = 20): received whole body vibration trained three times a week for 8 weeks

INTERVENTIONS:
Combination Product: Group A (n = 20): received core stability exercise trained three times a week for 8 weeks. — Woman was in crook lying position with feet flat on the treatment table. The therapist put his two thumbs on the anterior superior iliac spines then, asked the woman to contract the abdominal muscle, hold the contraction for 10 seconds, then, asked her to relax for 10 seconds
  Groups: Group A (n = 20): received core stability exercise trained three times a week for 8 weeks.
Device: Group B (n = 20): received whole body vibration trained three times a week for 8 weeks — The woman assumed a full squat position on a vibration platform. The apparatus was set at a frequency of 30 Hz, amplitude of 2 mm, and duration of 5 min. The women were instructed to remain in the squatting position with holding hand rail after turning on the vibration and to report any discomfort that might arise. At the end of 5 min, the vibration turned off automatically. Thereafter, the women took a 1-min rest. They were then asked to stand on the vibration platform for 5 min, with the same parameters as those used in the squatting position. Thus, the total time for the application of WBV in each session was 10 min
  Groups: Group B (n = 20): received whole body vibration trained three times a week for 8 weeks

SUMMARY:
This study was conducted to explore the influence of core stability exercise versus whole body vibration in improving vitamin D absorption in women.

DETAILED DESCRIPTION:
This study was conducted to explore the influence of core stability exercise versus whole body vibration in improving vitamin D absorption in women.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D concentration was less than 12ng/ml and age between 20 and 50 years and Their BMI less than 30

Exclusion Criteria:

* Vitamin D concentration was greater than 20ng/ml, Their BMI greater than 30 and exhibited a history of significant medical diseases such as rheumatoid diseases, uncontrolled high blood pressure, serious heart or lung issues, chronic viral infections including herpes and hepatitis

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research was conducted at the Physical Therapy Department of Al-Zaytoonah University. Forty female patients who had vitamin D deficiency were enrolled in this study according to specific criteria: vitamin D concentration was preliminarily assessed based on the parathyroid hormone response so concentration of vitamin D and parathyroid hormone were measured pre- and post-two month's intervention. Vitamin D concentration was less than 12ng/ml and age between 20 and 50 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-06-09 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
vitamin D concentration | 8 weeks
  Vitamin D concentration was less than 12ng/ml
parathyroid hormone | 8 weeks
  parathyroid hormone were measured pre- and post-two months intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous ishak shehata kelini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No